CLINICAL TRIAL: NCT05537831
Title: Ultrasound Guided vs Landmark-based Hematoma Block in Distal Forearm Fractures
Brief Title: Ultrasound Guided Hematoma Block in Distal Forearm Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Paul Klawitter, Associate Profressor, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1954614
Record Dates: First submitted 2022-09-02; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Forearm Fracture
Keywords: Ultrasound; Hematoma block
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Intervention Group (Ultrasound) (Active Comparator): The ultrasound probe will be used for real-time needle and hematoma localization using the linear probe. The hematoma block will then be performed with aseptic technique. The skin will be prepped with chlorhexidine. A 20-gauge needle will be inserted in-plane into the hematoma site. A small amount of blood will be aspirated to confirm placement and 5-10 mL of 1% lidocaine will be infiltrated.
  Interventions: Device: Ultrasound
- Study Control Group (Landmark) (No Intervention): The ultrasound probe will be in place on the patient's arm to maintain single blinding of the study. The ultrasound machine will not be used for needle and hematoma localization. The hematoma block will then be performed with aseptic technique. The skin will be prepped with chlorhexidine. A 20-gauge needle will be inserted in-plane into the hematoma site. A small amount of blood will be aspirated to confirm placement and 5-10 mL of 1% lidocaine will be infiltrated.

INTERVENTIONS:
Device: Ultrasound — The ultrasound will be used to assist with the delivery of a hematoma block in patients with distal forearm fractures.
  Arms: Study Intervention Group (Ultrasound)

SUMMARY:
This is a randomized control trial comparing the efficacy of ultrasound (US) guided vs landmark-guided hematoma blocks on distal forearm fractures.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than and equal to seven years of age
* Patients with traumatic acute distal radius/ulnar fractures with displacement that require reduction and immobilization with splinting
* Patients that receive distal radius hematoma blocks, including those who require additional pain control adjuncts if pain control is not adequate

Exclusion Criteria:

* Prisoners
* Pregnant women
* Patients with altered mental status/have impaired decision-making capacity.
* Patients with allergies to amide anesthetics

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Pain relief from landmark versus ultrasound guided hematoma block | Change in pain score from before the hematoma block to immediately after the reduction/splinting of the forearm fracture
  Pain will be measured using a ten point Likert scale with zero designated as no pain and ten being the worst pain the patient can imagine. The higher score the worse the outcome.

IPD SHARING:
Plan to Share IPD: No